CLINICAL TRIAL: NCT04050813
Title: Efficacy of Flywheel Inertial Resistance Training in the Architecture and Function of the Hamstrings in Athletes with a History of Hamstring Muscle Injury
Brief Title: Efficacy of Flywheel Inertial Resistance Training in the Architecture and Function of the Hamstring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Córdoba (Other)
Collaborators: Instituto Oulton (Unknown)
Responsible Party: Principal Investigator, Matias Sampietro, Principal Investigator, Universidad Nacional de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSMI MSampietro Tesis
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hamstring Injury
Keywords: Hamstring Injury; Flywheel Inertial Resistance; Hamstring architecture; Ultrasound; Eccentric
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): The program is performed 2 times per week using resistance equipment in a physiotherapy clinic. Each session consists of on 2-legged loaded exercises for hamstring, quadriceps, gluteus maximun and core. The patients complete 3 or 4 sets in each exercise with a 2- to 3-minute rest between sets and a 5-minute rest period between the 4 exercises.
  The number of repetitions decreases, and load gradually increases, every week. The repetitions and loads are as follows: 3 set of 12-repetition maximum (12RM), in week 1 and 2; 3 set of 10 RM, in week 3 and 4; 4 set of 10RM, in weeks 5 and 6; and 4 set of 8RM, in weeks 7 to 8.
  Interventions: Behavioral: Exercises program for hamstring architecture and function
- Intervention (Experimental): Experimental: Inertial flywheel resistance training The program is performed 2 times per week using resistance equipment in a physiotherapy clinical. Inertial flywheel resistance is a type of strength training; which is based on the increasing demands on eccentric action (breaking) after a concentric action (acceleration), due to the inertial load caused during the return movement. The patients complete 16 repetition maximum (RM) with moment inertia 0.05 m² from week 1-2, 24 repetition maximum (RM) with moment inertia = 0.10 m² from week 3 to 4. 32 repetition maximum (RM) with moment inertia = 0.10 m² from week 5 to 6 and 32 repetition maximum (RM) with moment inertia = 0.13 m² in a flywheel hamstring curl devise.
  Interventions: Behavioral: Exercises program for hamstring architecture and function

INTERVENTIONS:
Behavioral: Exercises program for hamstring architecture and function — To assess the effectiveness of the inertial flywheel resistance program in the architecture and function of the hamstrings post structural hamstring injury

SUMMARY:
Investigate the efficacy of the inercial Flywheel training protocol in modifying the architecture and function of the hamstrings in patients with a history of structural muscle injury vs conventional training.

The researchers hypothesize that inercial Flywheel training protocol will be a useful strategy in the modification of the architecture and function of the hamstring in patients with a history of indirect structural muscle injury and decrease the recurrence.

DETAILED DESCRIPTION:
Randomized controlled intervention study

ELIGIBILITY:
Inclusion Criteria:

* Adults with history of structural muscle injuries type 3 of the Munich Consensus classification for muscular injuries, confirmed by imaging diagnosis no more than 2 years ago.
* The patient must have performed conventional medical and physiotherapy treatment
* Have Returned to their usual sporting activity
* With good mental health.

Exclusion Criteria:

* Suffer from a systemic pathology that could alter the healing biology of the muscle.
* Present other lesions in the muscular group of extrinsic characteristic or not encompassed within type 3 structural lesions such as, for example, proximal or distal insertion tendinopathy, use of semitendinous as anterior cruciate ligament graft.
* Prior knee or hip surgery.
* Having been infiltrated with platelet rich plasma in the posterior thigth region in the previus 3 months before startin the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Change in the architecture and morphology of the hamstring | 0 and 8 week
  To assess change in architecture and morphology of the hamstring at 8 week. It will be performed by a medical specialist in diagnostic imaging with a A GE Voluson 730 Expert model ultrasound machine , with 6-12 MHz linear transducer. Panoramic images of the long portion of the biceps femoris and semitendinosus will be taken from its proximal insertion, In each muscle, muscle thickness, fascicle length, penetration angle and physiological cross-sectional area will be evaluated.
Change in Maximun isometric strength | 0 and 8 week
  To assess change in maximum isometric strength of hamstring in Newton (N). It will be measured in 3 repetitions with a hand dynamometer at two knee flexion angles.
Change in Rate of force development | 0 and 8 week
  To assess change in rate of force development of hamstring in N/seg at 8 week. it will be measured in 3 repetitions with a hand dynamometer at two knee flexion angles.
Change in Maximun eccentric strength | 0 and 8 week
  To assess the maximum eccentric strength of hamstring in Newton (N) from basiline. It will be measured in 3 repetitions with a hand held dynamometer.

SECONDARY OUTCOMES:
Change in Oslo hamstring injury screening questionnaire | 0 and 8 week
  Self-administered questionnaire. The hamstring injury detection test will be carried out to assess the previous injury, symptoms, function and quality of life of these players with the "Oslo hamstring injury screening questionnaire" questionnaire.This tool is divided in 23 items within 5 categories: symptoms, discomfort, pain depending on daily activity, sports and quality of life for injuries in right or left hamstrings
Functional scale of the lower limb | In the week before the 1st session of the protocol
  Self-reported patient-specific outcome measure assess functional change, primarily in patients presenting with musculoskeletal disorders. Patients are asked to identify up to 3 important activities they are unable to perform or are having difficulty with as a result of their problem. In addition to identifying the activities, patients are asked to rate, on an 11-point scale, the current level of difficulty associated with each activity. Following the intervention, patients are asked again to rate the activities previously identified. the lower limb will be used in its version validated in Argentina
Adverse events | week 8
  To capture all adverse events and side effects that occurred after exercises protocol. Patients reported any changes or any symptoms. If a question was answered "yes", we asked for further comments To capture all adverse events and side effects that occurred after exercises protocol. Patients reported any changes or any symptoms. If a question was answered "yes", we asked for further comments
Adherence self-report questionnaire | week 8
  Patients were asked to choose one of six descriptions (from level 1 = perfect adherence to level 6 = nonadherence) to express exercise treatment at the end of the twelve weeks study period.
Maximum Hip Flexion Active Knee Extension (MHFAKE) Test | 0 and 8 week
  to assess change in amplitude of movement of the hamstring in degrees with inclinometer
Single leg bridge test. Change in resistance of hamstring | 0 and 8 week
  to assess the ability or resistance of the hamstring in repetition numbers
Change in Test of a 1RM eccentric | 0 and 8 week
  To assess the maximun eccentric repetition in a conventional hamstring leg curl in kg

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Campana, Phd, Study Director — Departments of Biomedical Physics - University of Cordoba Argentina
Locations (1):
- Oulton GyMed, Rehabilitación y Gimnasio de Salud, Córdoba, Córdoba Province, Argentina

IPD SHARING:
Plan to Share IPD: No